CLINICAL TRIAL: NCT02570685
Title: Psychosocial Benefits of Gratitude Journals: A Randomized Controlled Intervention Trial
Brief Title: Psychosocial Benefits of Gratitude Journals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Brenda O'Connell, Ms. Brenda O' Connell, B.A., University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GratitudeJournal2015
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Happiness
Keywords: Gratitude Intervention; positive emotion; friendships; positive psychology; life satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reflective Interpersonal Gratitude (Experimental): An interpersonal gratitude journal, designed to foster gratitude for one's existing social relationships, by writing and reflecting on people and positive daily encounters for which one is grateful.
  Interventions: Behavioral: Reflective Interpersonal Gratitude
- Reflective-Behavioral Gratitude (Experimental): An interpersonal gratitude journal, designed to foster gratitude for one's existing social relationships, by writing and reflecting on people and positive daily encounters for which one is grateful. In addition participants are asked to choose a friend express this gratitude to them at the end of each week.
  Interventions: Behavioral: Reflective-Behavioral Gratitude
- Neutral Control Journal (Active Comparator): Write about and reflect on things that occurred over the course of the day.
  Interventions: Behavioral: Neutral Control Journal

INTERVENTIONS:
Behavioral: Reflective Interpersonal Gratitude — Participants were given the following instructions in their journal: Writing is a great way to reflect on your daily events, helping to look back and focus on the good things in our lives. There are many things in our lives, big and small, which we might be grateful for. For the next three weeks, 3 times a week (9 days in total), reflect back on your day and think of the people you met and interacted with and are grateful for. Please write down in the space provided a number of positive social interactions over the day or friendships/relationships you are grateful for…..
  Arms: Reflective Interpersonal Gratitude
Behavioral: Reflective-Behavioral Gratitude — Participants were given the following identical instructions as the reflective journal in addition to this "At the end of each week, express this gratitude to a friend of your choice face-to-face or through e-mail, facebook, a kind note, tell him/her how much you appreciate something specific that he/she does and reflect on how your friend's reaction and how you feel."
  Arms: Reflective-Behavioral Gratitude
Behavioral: Neutral Control Journal — Writing is a great way to reflect on your daily events, helping to look back and reflect on our lives. For the next three weeks, 3 times a week (9 days in total), please write in the spaces provided things that happened during the day.
  Arms: Neutral Control Journal

SUMMARY:
This randomized controlled study will examine the effects of different interpersonal gratitude journals compared to a neutral control journal on psycho social outcomes.

DETAILED DESCRIPTION:
This randomized controlled study will examine the effect of a) a reflective interpersonal gratitude journal, and b) an reflective and behavioral interpersonal gratitude journal, versus (c) an active control journal, on life satisfaction and other secondary outcomes. Explanatory mechanisms will be tested utilizing the broaden-and-build theory of positive emotions. Participants will be randomly assigned to one of these three conditions with three week, one month and three month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* English language proficiency

Exclusion Criteria:

* under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in Satisfaction With Life Scale (SWLS). Diener, E. D., Emmons, R. A., Larsen, R. J., & Griffin, S. (1985). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in life satisfaction levels over the course of the intervention and follow-ups.

SECONDARY OUTCOMES:
National Institute of Health Social Relationships Companionship Scale which assess Friendship Quality and Loneliness. Cyranowski, J. M., Zill, N., Bode, R., Butt, Z., Kelly, M. A., Pilkonis, P. A., & Cella, D. (2013). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in social relationships over the course of the intervention and follow-ups.
The Gratitude Questionnaire-Six Item Form (GQ-6) McCullough, M. E., Emmons, R. A., & Tsang, J. (2002). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in gratitude levels over the course of the intervention and follow-ups.

OTHER OUTCOMES:
The Expression of Gratitude in Relationships Scale. Lambert, N. M., Clarke, M. S., Durtschi, J. A., Fincham, F. D., & Graham, S. M. (2010). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in levels of gratitude expression over the course of the intervention and follow-ups.
The Four- item Relationship Satisfaction Scale. Funk, J. L., & Rogge, R. D. (2007). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in relationship satisfaction levels over the course of the intervention and follow-ups.
Depressive symptoms: CES-D 10 (Center for Epidemiologic Studies Depression Scale 10 item scale) Short Form. Andresen, E. M., Malmgren, J. A., Carter, W. B., & Patrick, D. L. (1994). | Baseline, immediate post-intervention at three weeks,,1 month, 3 months
  Used to assess changes in depressive symptom levels over the course of the intervention and follow-ups.
Relationship closeness: Inclusion of other in the Self Scale Aron, A., Aron, E. N., & Smollan, D. (1992). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  Used to assess changes in relationship closeness over the course of the intervention and follow-ups.
Scale of Positive and Negative Experiences , can use the Positive Feelings/affect subscale Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi. D., Oishi, S., & Biswas-Diener, R. (2009). | Baseline, immediate post-intervention at three weeks,1 month, 3 months
  potential moderator

CONTACTS AND LOCATIONS:
Overall Officials: Brenda O' Connell, B.A, Principal Investigator — University of Limerick; Stephen Gallagher, PhD, Study Director — University of Limerick; Deirdre O'Shea, PhD, Study Director — University of Limerick
Locations (1):
- University of Limerick, Limerick, Munster, Ireland